CLINICAL TRIAL: NCT00873600
Title: A Randomized Controlled Trial of Outpatient Geriatric Evaluation and Management Among Older Patients With Breast and Colon Cancer
Brief Title: Outpatient Health Care Program for Older Patients Receiving Chemotherapy for Newly Diagnosed Breast Cancer or Colon Cancer
Status: Withdrawn | Type: Observational
Why Stopped: No accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Cynthia Owusu, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Other Study IDs: CASE4Y07; P30CA043703 (NIH); CASE4Y07 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer; Cognitive/Functional Effects; Colorectal Cancer; Psychosocial Effects of Cancer and Its Treatment
Keywords: cognitive/functional effects; psychosocial effects of cancer and its treatment; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; adenocarcinoma of the colon; stage I colon cancer; stage II colon cancer; stage III colon cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Colonic Neoplasms | interventions — Drug Therapy; Chemotherapy, Adjuvant; Mental Status and Dementia Tests; Psychiatric Rehabilitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: chemotherapy
Other: medical chart review
Other: questionnaire administration
Procedure: adjuvant therapy
Procedure: assessment of therapy complications
Procedure: cognitive assessment
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Gathering health information from older patients undergoing chemotherapy may help doctors plan better treatment and improve the quality of life for these patients.

PURPOSE: This randomized clinical trial is studying how well an outpatient health care program works for older patients receiving chemotherapy for newly diagnosed breast cancer or colon cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the effect of a 1-year geriatric evaluation and management (GEM) program on adherence to adjuvant chemotherapy (defined as tolerance and timely completion of planned dose) in patients with newly diagnosed breast or colon cancer.

Secondary

* Evaluate the effect of a 1-year GEM program on the health-related quality of life and functional, cognitive, and mental status of these patients.
* Evaluate the effect of a 1-year GEM program on 3-year disease-free survival of these patients.
* Compare the number of emergency room visits, acute hospitalizations, and associated Medicare costs within the first 12 months following randomization to a GEM program vs no program.

OUTLINE: Patients are stratified according to tumor site (breast vs colon). Patients are randomized to 1 of 2 arms.

* Arm I (intervention): Patients complete health-related quality-of-life (QOL) and comprehensive geriatric assessment questionnaires at baseline, within 30 days after chemotherapy or at 6 months, and then at 12-13 months to assess functional status (i.e., activities of daily living), comorbidity (i.e., medical problems), medications, mood and memory, nutrition, and social support from family members and friends. Patients receive a home visit from a social worker and visit the Senior Adult Oncology clinic within 1 month after the first course of chemotherapy. The clinic staff develops an individualized care plan for the patient and communicates the results of the assessment questionnaires and their recommendations (e.g., medication and/or specialty referrals) to the patient's primary care provider and oncologist. The staff meets weekly to monitor and update the patient care plan. Patients are followed in the Senior Adult Oncology clinic at least every 3 months for 1 year. Follow-up telephone calls and in-home visits are also conducted as needed. Patients are also assessed prior to each course of chemotherapy for toxicities related to the chemotherapy.
* Arm II (control): Patients complete a health-related QOL questionnaire at baseline, within 30 days after chemotherapy or at 6 months, and then at 12-13 months. Patients receive oncology and primary care by their usual health care providers.

After completion of the study intervention, patients' medical charts are reviewed periodically for up to 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma, including one of the following:

  * Breast cancer (female), meeting the following criteria:

    * Stage I-III (T1-4, N0-3, M0) disease
    * Has undergone complete surgical removal of invasive cancer by mastectomy or lumpectomy
    * Has undergone either sentinel lymph node dissection or axillary lymph node dissection with adequate TNM staging
  * Colon cancer (male or female), meeting the following criteria:

    * Stage I-III (T1-3, any N, M0) disease
    * Has undergone appropriate surgical resection with TNM staging
* Newly diagnosed disease
* Scheduled to receive chemotherapy

  * Agrees to receive chemotherapy AND is able to receive chemotherapy within 3 months after surgery
* No distant metastases
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Life expectancy ≥ 6 months
* Fluent in English
* Not living in a nursing home
* No end-stage disease
* No severe dementia
* No other clinically active malignancy within the past 5 years or within 3 months after diagnosis of current malignancy

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy for the malignancy
* More than 1 year since prior treatment on an inpatient/outpatient geriatric evaluation and management unit

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-10

PRIMARY OUTCOMES:
Chemotherapy tolerability as measured by dose reduction, treatment delay, and incidence of grade 3-5 toxicities

SECONDARY OUTCOMES:
Mean change in comprehensive geriatric assessment scores and quality-of-life scores from baseline to post-chemotherapy and from baseline to 12 months following randomization
Number of emergency room visits, acute hospitalizations, and associated Medicare costs within the first 12 months following randomization
3-year disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Owusu, MD, MSC, Principal Investigator — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://clinicaltrials.gov/ct2/results?term=case4y07